CLINICAL TRIAL: NCT01288898
Title: A Double-blind, Placebo-controlled, Dose Escalating Study to Assess the Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of ASP1941 and to Explore the Effect of ASP1941 on Urine and Blood Glucose Levels in Healthy Subjects
Brief Title: Multiple Dose Escalating Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP1941
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 1941-CL-0002; 2006-006525-11 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: ASP1941; Diabetes Mellitus; Multiple ascending doses; Healthy subjects
MeSH Terms: conditions — Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ASP1941 — Oral
Drug: Placebo — Oral

SUMMARY:
This study determined the safety of ASP1941 after a single and multiple once-daily doses for 10 days in healthy subjects. In addition, the Pharmacokinetics (PK) and Pharmacodynamics (PD) of ASP1941 were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60-100kg, body mass index (BMI) between 20-30 kg/m2, inclusive

Exclusion Criteria:

* Fasting Plasma Glucose (FPG) > 6.4 mmol/l
* HbA1c > 6.2%
* Abnormal pulse of blood pressure at screening, as judged by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability assessed by the incidence of adverse events, vital signs, physical examinations, 12-lead ECG and lab-tests | 31 days

SECONDARY OUTCOMES:
Pharmacokinetics assessed by the ASP1941 plasma concentration change | up to 96 hours after last dose
Pharmacodynamics assessed by the ASP1941 glucose concentration changes in blood and urine | up to 96 hours after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Groningen, Netherlands

REFERENCES:
- [Derived] Veltkamp SA, Kadokura T, Krauwinkel WJ, Smulders RA. Effect of Ipragliflozin (ASP1941), a novel selective sodium-dependent glucose co-transporter 2 inhibitor, on urinary glucose excretion in healthy subjects. Clin Drug Investig. 2011 Dec 1;31(12):839-51. doi: 10.1007/BF03256922. PMID 21877761